CLINICAL TRIAL: NCT06221826
Title: Prospective Randomized Study of the Modulating Effect of MEXIDOL® as an Adjuvant Stimulant of the Cognitive-emotional Component of the Rehabilitation Treatment in Patients With Acute Cerebral Failure
Brief Title: MEXIDOL® in the Rehabilitation Treatment of Patients With Acute Cerebral Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pharmasoft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MexidolNeuro2023
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke; Acute Stroke; Cerebral stroke; Traumatic Brain Injury; Acute Cerebrovascular Accident; ACVA; Acute cerebral failure; Neuroprotection; Mexidol; Ethylmethylhydroxypyridine Succinate
MeSH Terms: conditions — Ischemic Stroke; Stroke; Brain Injuries, Traumatic | interventions — emoxypine succinate; ethylmethylhydroxypyridine succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main (Mexidol and standard treatment) (Experimental): Mexidol IV 500 mg for 10 days, then Mexidol FORTE 250 orally 250 mg 1 tablet 3 times a day for 8 weeks; and standard treatment
  Interventions: Drug: Mexidol
- Control (No Intervention): Standard treatment: basic practices of kinesitherapy, occupational therapy, speech therapy, clinical psychology, supplemented by adjuvant procedures of electrotherapy and rehabilitation environment therapy. The patient's rehabilitation load was at least 3 hours a day for 12 days

INTERVENTIONS:
Drug: Mexidol — Neurocytoprotector
  Other Names: Ethylmethylhydroxypyridine Succinate
  Arms: Main (Mexidol and standard treatment)

SUMMARY:
The use of metabolic modulators creates prospects for increasing the efficiency of the rehabilitation treatment of patients with acute cerebral failure

DETAILED DESCRIPTION:
Modern neurorehabilitation is a set of basic and adjuvant treatment methods that provide a modulating effect on the neurorestoration process. The range of basic rehabilitation practices includes kinesiotherapy, occupational therapy, speech therapy, and neuropsychology. Adjuvant methods include physiotherapeutic and medicinal methods. For this study, the investigators chose MEXIDOL® as an adjuvant metabolic medicine, which has the ability to modulate receptor complexes of brain membranes, in particular benzodiazepine, GABA, acetylcholine, enhancing their ability to bind to specific ligands. This pharmacodynamic feature of the drug can have a positive effect on the psycho-emotional state of patients, which in turn will increase motivation and, consequently, the success of the rehabilitation process

ELIGIBILITY:
Inclusion Criteria:

* Acute Ischemic Stroke
* Montreal Cognitive Assessment (MoCA) test >15; ≤22

Exclusion Criteria:

* Under 18 years old
* Epilepsy
* Pregnancy
* Acute failure of one or more organ systems
* Purulent-inflammatory disease of any localization
* Participating in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Institute Clinic, Yekaterinburg, Sverdlovsk Oblast, Russia

REFERENCES:
- [Background] Belkin AA, Belkin VA, Vasilchenko IE, Pinchuk EA. [Results of a cohort single-center randomized study of the modulating effect of the drug Mexidol in the rehabilitation of patients who suffered acute cerebral insufficiency]. Zh Nevrol Psikhiatr Im S S Korsakova. 2024;124(4):108-117. doi: 10.17116/jnevro2024124041108. Russian. PMID 38676685
- See also: Belkin AA, Belkin VA, Vasilchenko IE, Pinchuk EA. [Results of a cohort single-center randomized study of the modulating effect of the drug Mexidol in the rehabilitation of patients who suffered acute cerebral insufficiency] — https://www.mediasphera.ru/issues/zhurnal-nevrologii-i-psikhiatrii-im-s-s-korsakova/2024/4/1199772982024041108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Main (Mexidol and Standard Treatment) | Control | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 6 | 31
  >=65 years | 5 | 24 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (10.3) | 66.6 (9.4) | 65.3 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 17 | 30
  Male | 17 | 13 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 30 | 30 | 60
Cognitive status [MoCA] [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA test) [31 point scale: min value 0, max value 30, higher scores mean a better outcome]
  units on a scale | 19.1 (2.26) | 19.6 (1.83) | 19.35 (2.05)
The Rehabilitation Routing Scale (RRS) [Mean (Standard Deviation); unit: units on a scale] — The Rehabilitation Routing Scale (RRS) [7 point scale: min value 0, max value 6, higher scores mean a worse outcome]
  units on a scale | 3.9 (0.4) | 4.1 (0.5) | 4.0 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Аssessment of Attentiveness and Performance
Description: Schulte test [work efficiency]. Test methodology: the subject is successively shown 5 tables (5x5), in the cells of which numbers (from 1 to 25) are randomly located. It is required to show and name all the numbers in ascending order (from 1 to 25). The time spent on each table separately is recorded. Depending on the objectives, the excess of the standard (40-50 sec) time spent on each table and the dynamics of time indicators, or the average or total result of the examination for all five tables, are analyzed [test time: min value 30.0 sec, max value N/A; higher scores mean a worse outcome].
Time Frame: Assessed before starting therapy (Day 1), at the end of the parenteral therapy phase (Day 10) and at the end of the course of therapy (Day 66).
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
seconds
  Day 1 | 94.9 [69.35 to 114.95] | 71.2 [65.15 to 87.9]
  Day 10 | 75 [60.9 to 95.7] | 68.15 [62.15 to 88.65]
  Day 66 | 71.7 [56.65 to 102.3] | 63 [55.73 to 82.95]

2. Primary Outcome: Dynamics of Cognitive Status
Description: The Montreal Cognitive Assessment (MoCA test) [31 point scale: min value 0, max value 30, higher scores mean a better outcome]
Time Frame: Assessed at screening (Day 0), at the end of the parenteral therapy phase (Day 10) and at the end of the course of therapy (Day 66); Day 66 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 23.8 (2.6) | 22.9 (3.0)

3. Primary Outcome: Severity of Depression
Description: The Beck Depression Inventory (BDI scale) [64 point scale: min value 0, max value 63, higher scores mean a worse outcome]
Time Frame: Assessed before starting therapy (Day 1), at the end of the parenteral therapy phase (Day 10), in the middle of the oral therapy phase (Day 38) and at the end of the course of therapy (Day 66); Day 66 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 7.5 (4.5) | 11.4 (5.6)

4. Primary Outcome: Reduction in Anxiety
Description: The Hospital Anxiety and Depression Scale (HADS) [22 point scale: min value 0, max value 21, higher scores mean a worse outcome]
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 2.6 (2.4) | 4.4 (2.4)

5. Primary Outcome: Severity of Post Intensive Care Syndrome
Description: The Post Intensive Care Syndrome (PICS) score [21 point scale: min value 0, max value 10 with 0,5 point scale division, higher scores mean a worse outcome]
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 0.02 (0.09) | 0.3 (0.6)

6. Primary Outcome: Dynamics of Level of Mobility
Description: The Rivermead index [16 point scale: min value 0, max value 15, higher scores mean a better outcome]
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 10.3 (2.8) | 8.0 (2.8)

7. Primary Outcome: Dynamics of the Level of Life
Description: The Rehabilitation Routing Scale (RRS) [7 point scale: min value 0, max value 6, higher scores mean a worse outcome]
Time Frame: Assessed at screening (Day 0), at the end of the parenteral therapy phase (Day 10), in the middle of the oral therapy phase (Day 38) and at the end of the course of therapy (Day 66); Day 66 reported
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 2.9 (0.7) | 3.3 (0.6)

8. Primary Outcome: Severity and Dynamics of Muscle Strength
Description: The Muscle Strength Quantitative Rating (MRC) Scale [6 point scale: min value 0, max value 5, higher scores mean a better outcome]
Time Frame: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
score on a scale | 3.3 (5.1) | 2.1 (2.2)

9. Primary Outcome: Systolic Cerebral Blood Flow Velocity (Vs) Using Transcranial Doppler (TCD) at Key Time Points
Description: Systolic cerebral blood flow velocity (Vs) was measured in сm/sec using transcranial Doppler ultrasonography (TCD). Measurements were taken for each participant at five key time points: (1) before the first Mexidol infusion ("Before infusion"), (2) at the start of the infusion, (3) at the start of the Schulte test, (4) at the end of the Schulte test, and (5) at the end of the infusion. [Normal values: min 35 сm/sec, max 95 сm/sec]
Time Frame: The TCDG parameters registrated before infusion, at the start of the infusion, at the start of the Schulte test, at the end of the Schulte test, at the end of the infusion.
Measure: Mean (Standard Deviation); unit: сm/sec
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
сm/sec
  Before infusion | 72.6 (18.41) | 80.03 (33.49)
  Start of the infusion | 72.23 (17.68) | 80.8 (33.09)
  Start of the Schulte test | 74.6 (18.73) | 83.57 (34.3)
  End of the Schulte test | 76.83 (17.76) | 80.87 (31.98)
  End of the infusion | 78.53 (17.78) | 83.57 (32.29)

10. Primary Outcome: Overshoot Coefficient (OC) of Systolic Cerebral Blood Flow Velocity (TCD) at Key Time Points
Description: The Overshoot Coefficient (OC) is a ratio reflecting the change in systolic cerebral blood flow velocity before and after specific stimuli. It was calculated based on transcranial Doppler measurements at five key time points: (1) before the first Mexidol infusion ("Before infusion"), (2) at the start of the infusion, (3) at the start of the Schulte test, (4) at the end of the Schulte test, and (5) at the end of the infusion. [It's calculated by the formula OC=(Vo-Vs)/Vs, the norm is not less than 1.12]
Time Frame: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
ratio
  Before infusion | 1.25 (0.05) | 1.27 (0.05)
  Start of the infusion | 1.26 (0.04) | 1.27 (0.04)
  Start of the Schulte test | 1.25 (0.05) | 1.27 (0.04)
  End of the Schulte test | 1.26 (0.05) | 1.27 (0.04)
  End of the infusion | 1.27 (0.05) | 1.28 (0.04)

11. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Registration of adverse events related to Mexidol and significant differences in vital signs between groups
Time Frame: Throughout the study [From Day 1 up to Day 66]
Measure: Number; unit: Adverse events
Arm/Group | Main (Mexidol and Standard Treatment) | Control
Number analyzed (Participants) | 30 | 30
Adverse events | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout the study [From Day 1 up to Day 66]
Description: No adverse events were reported in the study
Arm/Group | Main (Mexidol and Standard Treatment) | Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT06221826/Prot_SAP_000.pdf